CLINICAL TRIAL: NCT00389922
Title: Phase I Study of Two Different Schedules of Lapatinib (GW572016) in Combination With Vinorelbine in Advanced Solid Tumors
Brief Title: Lapatinib and Vinorelbine in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000505878; P30CA093373 (NIH); UCDCC-171 (Other: University of California, Davis - Cancer Center); UCDCC-200513681-1 (Other: University of California, Davis - IRB); GSK-104241 (Other: GlaxoSmithKline)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Lapatinib; Vinorelbine; Comparative Genomic Hybridization; Cytogenetic Analysis; Gene Expression Profiling; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis; Reverse Transcriptase Polymerase Chain Reaction; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Daily Dosing) (Experimental): Oral lapatinib given daily for 28 days plus IV vinorelbine given weekly (3 out of 4 weeks)
  Cohorts of 3-6 patients receive escalating doses of lapatinib ditosylate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity during course 1. At least 6 patients are treated at the MTD. Once the MTD of lapatinib has been determined, patients may be accrued to group B or to a separate pharmacokinetics cohort in group A.
  Interventions: Drug: lapatinib ditosylate; Drug: vinorelbine ditartrate; Genetic: comparative genomic hybridization; Genetic: cytogenetic analysis; Genetic: gene expression analysis; Genetic: mutation analysis; Genetic: polymerase chain reaction; Genetic: polymorphism analysis; Genetic: proteomic profiling; Genetic: reverse transcriptase-polymerase chain reaction; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis
- B (Intermittent Dosing) (Experimental): Oral lapatinib given days 2-5, 9-12 and 16-25 plus IV vinorelbine given weekly (3 out of 4 weeks)
  Cohorts of 3-6 patients receive escalating doses of lapatinib ditosylate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity during course 1. At least 6 patients are treated at the MTD. Once the MTD of lapatinib has been determined, patients may be accrued to group B or to a separate pharmacokinetics cohort in group A.
  Interventions: Drug: lapatinib ditosylate; Drug: Vinorelbine ditartrate

INTERVENTIONS:
Drug: lapatinib ditosylate — Given orally for 28 days per dose level (Dose level 1: 250mg; Dose level 2: 500mg; Dose level 3: 1000mg; Dose level 4: 1250mg; Dose level 5: 1500mg; Dose level 6: 1500mg)
  Other Names: Tykerb
  Arms: A (Daily Dosing)
Drug: vinorelbine ditartrate — Given IV Days 1, 8 and 15 per dose level (Dose level 1: 20mg/m2; Dose level 2: 20mg/m2; Dose level 3: 20mg/m2; Dose level 4: 20mg/m2; Dose level 5: 20mg/m2; Dose level 6: 25mg/m2)
  Other Names: Navelbine
  Arms: A (Daily Dosing)
Genetic: comparative genomic hybridization — Molecular correlative study
  Arms: A (Daily Dosing)
Genetic: cytogenetic analysis — Molecular correlative study
  Arms: A (Daily Dosing)
Genetic: gene expression analysis — Molecular correlative study
  Arms: A (Daily Dosing)
Genetic: mutation analysis — Molecular correlative study
  Arms: A (Daily Dosing)
Genetic: polymerase chain reaction — Molecular correlative study
  Arms: A (Daily Dosing)
Genetic: polymorphism analysis — Molecular correlative study
  Arms: A (Daily Dosing)
Genetic: proteomic profiling — Molecular correlative study
  Arms: A (Daily Dosing)
Genetic: reverse transcriptase-polymerase chain reaction — Molecular correlative study
  Arms: A (Daily Dosing)
Other: immunohistochemistry staining method — Molecular correlative study
  Arms: A (Daily Dosing)
Other: laboratory biomarker analysis — Molecular correlative study
  Arms: A (Daily Dosing)
Drug: lapatinib ditosylate — Given orally on Days 2-5, 9-12 and 16-25 per dose level (Dose level 1: 1250mg; Dose level 2: 1500mg; Dose level 3: 1500mg; Dose level 4: 1700mg)
  Other Names: Tykerb
  Arms: B (Intermittent Dosing)
Drug: Vinorelbine ditartrate — Given IV Days 1, 8 and 15 per dose level (Dose level 1: 20mg/m2; Dose level 2: 20mg/m2; Dose level 3: 25mg/m2; Dose level 4: 25mg/m2)
  Other Names: Navelbine
  Arms: B (Intermittent Dosing)

SUMMARY:
RATIONALE: Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as vinorelbine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving lapatinib together with vinorelbine may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of lapatinib when given together with vinorelbine in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of 2 different schedules of lapatinib ditosylate when administered with vinorelbine ditartrate in patients with advanced solid tumors.

Secondary

* Determine the maximum tolerated dose (MTD) of each of these regimens in these patients.
* Determine, preliminarily, the efficacy of these regimens in these patients.
* Examine tissue and blood specimens from these patients to investigate potential predictors of response.
* Determine the pharmacokinetics of lapatinib ditosylate and vinorelbine ditartrate in patients treated at the MTD.

OUTLINE: This is a phase I study comprising 2 separate, sequential dose-escalation studies of lapatinib ditosylate. Patients are assigned to 1 of 2 treatment groups.

* Group A (daily dosing): Patients receive oral lapatinib ditosylate once daily on days 1-28 and vinorelbine ditartrate IV on days 1, 8, and 15.

Cohorts of 3-6 patients receive escalating doses of lapatinib ditosylate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity during course 1. At least 6 patients are treated at the MTD. Once the MTD of lapatinib has been determined, patients may be accrued to group B or to a separate pharmacokinetics cohort in group A.

* Pharmacokinetics (PK) cohort*: Patients in the PK cohort receive vinorelbine ditartrate IV as in group A and oral lapatinib ditosylate once daily at the MTD on days 3-28 (course 1 only) and on days 1-28 in all subsequent courses. Patients undergo PK sampling during course 1.

NOTE: *Accrual to group B and to the PK cohort of group A may occur simultaneously.

* Group B (intermittent dosing): Patients receive oral lapatinib ditosylate once daily at the MTD on days 2-5, 9-12, and 16-25 and vinorelbine ditartrate IV, on days 1, 8, and 15.

In both groups and in the PK cohort, treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients who have completed 6 courses of combined therapy may receive additional courses with lapatinib ditosylate alone.

Patients undergo blood collection and buccal brushings periodically for pharmacokinetic and biomarker correlative studies. Archival tumor tissue is also evaluated for biomarkers, including epidermal growth factor receptor (EGFR) and HER-2/neu expression levels, EGFR polymorphisms and gene mutations (including RAS), levels of cellular proliferation and apoptosis, and RAS mutations by immunohistochemistry, mutation analysis, TUNEL assay, and polymerase chain reaction.

After completion of study treatment, patients are followed for 30 days.

PROJECTED ACCRUAL: A total of 66 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically proven advanced solid tumors for which there is no known standard therapy available or are not eligible for standard therapy because of their performance status, or have progressed after no more than 2 prior chemotherapy regimens for metastatic disease.
* Measurable or evaluable disease. Disease in previously irradiated sites is considered measurable if there is clear disease progression following radiation therapy.
* 18 years of age or older.
* Zubrod performance status of 0-2.
* Estimated survival of at least 3 months.
* Any prior chemotherapy must have been completed at least 4 weeks prior to start of this protocol and all side effects (except alopecia) resolved to grade 1 or less. Any prior radiation must have been completed at least 2 weeks prior to start of therapy. For prior mitomycin chemotherapy a 6-week interval is required. Patients must have completed prior trastuzumab at least 4 weeks prior to start of protocol therapy.
* Adequate renal function
* Adequate liver function
* Pretreatment granulocyte count of >1500/mm3 and platelet count of >100 000/mm3.
* Cardiac ejection fraction within the institutional range of normal as measured by 2-D echocardiogram or MUGA scan.
* Asymptomatic treated brain metastasis may be included if they are neurologically stable and have been off steroids and anticonvulsants for at least 4 weeks.
* All patients must give informed consent.
* Able to take and retain oral medication.
* Patients of reproductive potential must agree to use an effective contraceptive method

Exclusion Criteria:

* Patients may not have previously received lapatinib, vinorelbine or any other EGFR-1 targeted agent. Prior trastuzumab is allowed.
* Females cannot be pregnant or breastfeeding
* Symptomatic brain metastasis or still requiring steroids and anticonvulsants may not participate.
* Pre-existing neuropathy > grade 2 may not participate.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, will be excluded.
* History of other diseases, metabolic dysfunction, physical examination finding or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the patient at high risk from treatment complications.
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, or prior surgical procedures affecting absorption.
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with lapatinib.
* Patients requiring oral anticoagulants are eligible provided there is appropriate close INR monitoring is in place. If medically appropriate and treatment available, the investigator may also consider switching these patients to LMW heparin, where an interaction with lapatinib is not expected.
* Adherence to the requirements for concomitant medications classified as CYP3A4 inducers or inhibitors, or gastric pH modifiers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-12; Primary Completion 2009-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Toxicity as assessed by NCI CTCAE v3.0 | Completion of study

SECONDARY OUTCOMES:
Maximum tolerated dose of lapatinib ditosylate when administered with vinorelbine ditartrate as assessed by NCI CTCAE v3.0 | Completion of study
Response rate (complete response, partial response, progressive disease, and stable disease) assessed at baseline and prior to courses 3 and 5 | Completion of study
Best response | Completion of study
Survival | Completion of study
Progression-free survival | Completion of study
Biological markers as predictors of response | Completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Helen K. Chew, MD, Study Chair — University of California, Davis
Locations (4):
- United States (4):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - Seattle Cancer Care Alliance, Seattle, Washington